CLINICAL TRIAL: NCT03455010
Title: Dose-Response Relationship of Ambulatory Load and Cartilage - Pilot Study
Acronym: COMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Erlangen-Nürnberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-01006
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: Ambulatory load; Biomarker; Articular cartilage

STUDY DESIGN:
Intervention Model Description: Controlled multimodal data collection (biological, biomechanical) with block randomization.
Masking Description: Masking is not possible because the experimental condition is obvious. Participants and testers cannot influence outcome parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal load (No Intervention): Healthy subjects walking for 30 minutes on a treadmill with normal body weight
- Increased load (Experimental): Healthy subjects walking for 30 minutes on a treadmill with 20% additional body weight
  Interventions: Other: Increased load
- Reduced load (Experimental): Healthy subjects walking for 30 minutes on a treadmill with 20% lower body weight
  Interventions: Other: Reduced load

INTERVENTIONS:
Other: Increased load — Participants walk with 120% body weight achieved with a weight vest
  Arms: Increased load
Other: Reduced load — Participants walk with 80% body weight achieved by a dynamic unloading system
  Arms: Reduced load

SUMMARY:
The research question is if there is a dose-response relationship between blood biomarkers for articular cartilage and the magnitude of physiological load. To investigate this load induced biomarker change, the participants will complete a 30-minute walking test under three loading conditions: A: 80%, B: 100% C: 120% of their respective bodyweight (Fig. 1).

The main biomarker we are interested in is called cartilage oligomeric matrix protein (COMP). Serum COMP levels are increased immediately after 30-min running but there is no dose-response relationship shown yet.

DETAILED DESCRIPTION:
The current state of research in the field and of our own research clearly shows that the in vivo mechanobiology of articular cartilage is poorly understood. Previous results of changes in cartilage biomarker concentrations after ambulatory exercise raise the following question:

Do load-induced changes in blood biomarkers for articular cartilage (COMP) depend on the physiological load magnitude? To generate initial data for answering this question, we will establish the experimental framework to systematically study the in vivo mechanobiology of human articular cartilage to address the following aims.

* To obtain pilot data for investigating the in vivo dose-response relationship of weight-bearing and blood levels of mechanosensitive biomarker of articular cartilage using controlled load- bearing as experimental paradigm.
* To provide pilot data for comparing ambulatory biomechanics between the controlled load- bearing conditions.

The experimental setting consists of a 30-minutes walking stress test under three loading conditions: A: 80 %, B: 100% and C: 120% bodyweight. Unloading will be achieved through an unloading system and additional loading with an adjustable weight vest. Before and after the walking stress test, venous blood samples will be taken at five time points. The biomarker concentration is measured with a commercial available enzyme-linked immunosorbent assay (ELISA).

Hypothesis Our working hypothesis is that there is a dose-response relationship between the temporarily increased or decreased load and the load-induced change in COMP level in the blood serum. We assume that serum COMP concentration increases with increasing accumulated load on the knee cartilage simulated through the three different loading conditions.

Design The design of the pilot study is a controlled multimodal data collection (biological, biomechanical) with block randomization. Specifically, we will collect blood samples and biomechanical (kinematic and pressure) data. We will determine the relationship between the serum blood concentration and the biomechanical data.

Because this is a cross-over study, all participants will perform the same three walking stress tests but in random order. Each participant of the study will be tested for 2.5 hours on 3 separate days.

Method In this experiment, we will test 24 healthy participants (12 male, 12 female) on 3 test days under three different loading conditions in a randomized block design. On each test day, participants will complete walking stress test for 30-minutes with A: 80%, B: 100% and C: 120% of their bodyweight. Through the modified bodyweight we generate higher or lower forces on the knee cartilage, which should affect the COMP concentration in the blood serum.

To measure the change in serum COMP concentration, blood samples will be taken at five time points before and after the walking stress test. The blood samples are taken by a study nurse. For the venipuncture, a thin, sterile, disposable vein catheter is placed in the antecubital vein. The catheter stays in the vein for the entire 2.5 hours of the experiment. Blood samples will be collected and allowed to clot for 30-minutes. Serum will be separated and frozen in aliquots to -20°C within 1 hour of collection and then transferred for storage at -80°C until assayed. Serum biomarker concentrations will be determined using commercial ELISAs.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* being physically active (> 2/week)
* body mass index (BMI) <30 kg/m2

Exclusion Criteria:

* previous knee injury
* neuromuscular condition affecting gait

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Load-induced serum Cartilage Oligomeric Matrix Protein concentration | 3 hours
  Change in serum concentration during 30-minute walking exercise determined by commercial ELISA 30 min before to 2 hours after 30-minute walking exercise

SECONDARY OUTCOMES:
Overall ground reaction force impulse | 30 minutes
  Area under the ground reaction curve multiplied by number of steps taken during 30-minute walking exercise
Dynamic range of motion lower extremity joints | 30 minutes
  Min to max joint angles (ankle, knee, hip) measured using RehaGait (inertial measurement units)

OTHER OUTCOMES:
Age | At enrollment
  Age in years
Sex | At enrollment
  male or female
Body mass index | At enrollment
  BMI in kg/m2
Knee function | At enrollment
  Knee Osteoarthritis Outcome Score measured by questionnaire (best score: 100 - no limitations; worst score: 0)

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Muendermann, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No